CLINICAL TRIAL: NCT06500494
Title: Advanced Breast Cancer Patients Treated With Oral Vinorelbine: a Prospective and Retrospective, Observational Study - VINOREAL
Brief Title: To Describe How Well Vinorelbine Given Orally Works in Patients With a Breast Cancer After 2 Years of Treatment
Acronym: VINOREAL
Status: Recruiting | Type: Observational
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS16760
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Vinorelbine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: Patients who initiated an oral vinorelbine treatment for advanced breast cancer over the 2011-2020 targeted enrollment period
  Interventions: Drug: Vinorelbine Tartrate Oral
- Prospective Cohort: Patients initiating an oral vinorelbine treatment for advanced breast cancer at or after inclusion in the study and eligible for prospective collection of QoL data and PPQ and WPAI questionnaires
  Interventions: Drug: Vinorelbine Tartrate Oral

INTERVENTIONS:
Drug: Vinorelbine Tartrate Oral — The recommended dosage for oral vinorelbine is 60 mg/m² of body surface area (BSA) administered once weekly for the first three weeks, followed by 80 mg/m² of BSA for the following weekly administration.
  Other Names: Navelbine

SUMMARY:
This study looks at how well oral vinorelbine works in treating advanced breast cancer. It looks at women who have already had this treatment or are currently having it.

DETAILED DESCRIPTION:
This is an international, multicenter, retrospective and prospective, observational study.

The study will comprise of two cohorts:

* Retrospective: Patients who started OV treatment for ABC between 2011 and 2020 will be enrolled in the retrospective cohort study. The observation period for retrospectively included patients will extend from the initiation of OV treatment to the date of death, date of last contact or end date of retrospective observation period, whichever occurs first. The end date of retrospective observation period will be set as the date of the inclusion of the first patient in the study (First Patient In= FPI).
* Prospective: Patients initiating OV treatment and eligible for prospective collection of QoL data and PPQ and WPAI questionnaires will be enrolled in the prospective cohort study. The enrollment period is expected to extend up to 17 months from study start. The study observation period will extend up to 2 years after last patient first visit (around 24 months after treatment initiation).

Due to the observational nature of this study, no additional medical procedures or in person clinical visits beyond routine oncology care will be required for this study.

ELIGIBILITY:
Inclusion Criteria:

Female aged ≥ 18 years (≥ 19 years for Algeria as per local regulation) at oral vinorelbine ( OV) -based treatment initiation

Confirmed diagnosis of locally advanced or metastatic breast cancer eligible for chemotherapy

Initiated OV-based treatment as per SmPC for advanced breast cancer between January 2011 and December 2020 for the retrospective cohort or, initiating oral vinorelbine treatment at enrollment for the prospective cohort

Willing and able to complete the QoL questionnaire, PPQ and WPAI questionnaire for the prospective cohort

Provision of informed consent or non-opposition to the patient (or next of kin/legal representative, if applicable) for the use of data, according to local regulations

Exclusion Criteria:

no exclusion criteria for patients in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Study Population: The study population will include advanced breast cancer (ABC) patients treated with Oral Vinorelbine in any line of treatment and living in one of the target countries (Italy, China and Algeria).
  ABC includes locally advanced breast cancer and metastatic breast cancer either newly diagnosed or a relapse.
  The retrospective cohort will include 130 patients who initiated oral vinorelbine-based therapy (OV) in any line of treatment between 2011 and 2020, whether they are alive, have progressed or have died by the time of data collection.
  The prospective cohort will include 238 patients for whom it is planned, at the time of study enrollment, to receive oral vinorelbine in any line of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
PFS rate in both cohorts. | 2-years follow-up
  PFS is defined as the time between vinorelbine-based treatment initiation and the first occurrence of progression or death from any cause, with censoring of patients who are lost to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Eric Garrigue, MD, Study Chair — Pierre Fabre Medicament
Locations (3):
- Centre Hospitalo-Universitaire Mustapha, Hopital Mustapha, Place du 1er Mai 1945, Sidi M'Hamed, Algiers, Algeria
- Tianjing Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China
- Azienda Ospedaliera San Gerardo U.O. Oncologia Medica, Monza, Italy

IPD SHARING:
Plan to Share IPD: No